CLINICAL TRIAL: NCT07063654
Title: Creating a Mobile Health Program for Teens With Congenital Heart Disease
Brief Title: Mobile Health Program for Teens With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristen Fox (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Kristen Fox, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003377; K23HL166771 (NIH)
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Congenital Heart Disease in Adolescence; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Health Program (Experimental): Participants in this arm will receive access to Heart2Heart. Heart2Heart is a mobile health program for teens with congenital heart disease. It includes information and interactive features to help teens learn about staying healthy with congenital heart disease.
  Interventions: Behavioral: Heart2Heart

INTERVENTIONS:
Behavioral: Heart2Heart — Heart2Heart is a mobile health program for teens with congenital heart disease. It includes information and interactive features to help teens learn about staying healthy with congenital heart disease.

SUMMARY:
The goal of this clinical trial is to understand what teens with congenital heart disease like and want in a mobile health program that helps them learn about their health and make healthy choices. The main questions it aims to answer are:

Are participants satisfied with the program? Is the program easy to use?

Participants will: 1) complete two online surveys, 2) interact with the mobile health program, and 3) participate in an interview.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of structural congenital heart disease
* 12-18 years of age at time of study enrollment

Exclusion Criteria:

* Cognitive impairments limiting the ability to complete surveys or interviews
* Not proficient in the English language
* Leaving the United States during the study period

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2025-07-17 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Satisfaction with mHealth Program | Two weeks after receiving access to the mobile health program
  Participants' satisfaction with the mobile health program, for example, how much it increased their knowledge and how enjoyable it was. Participants respond to questions on a 4-point scale ("Strongly Disagree to Strongly Agree").
Usability of mHealth Program | Two weeks after receiving access to the mobile health program
  How easy and enjoyable participants think the program is to use, for example, how easy it was to find information or how much they liked the images. Participants respond to questions on a 7-point scale (1="Very Unsatisfied", 7="Very Satisfied").

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No